CLINICAL TRIAL: NCT02784782
Title: Thoracolumbar Burstfractures, Orthesis or no Orthesis
Acronym: BONO
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Elisabeth-TweeSteden Ziekenhuis (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Principal Investigator, Wouter Bakker, drs., Elisabeth-TweeSteden Ziekenhuis
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ElisabethTweeStedenZ
Record Dates: First submitted 2016-03-15; First posted 2016-05-27 (Estimated); Last update posted 2016-05-27 (Estimated); Status verified 2016-05

CONDITIONS: Spinal Fractures
Keywords: Spinal; Vertebral; Burstfracture; Orthesis; Brace; Thoracolumbar
MeSH Terms: conditions — Spinal Fractures | interventions — Functional Status

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Orthesis (Experimental): Subjects will wear a TLSO for 6 weeks 24 hours a day or they will not. After 6 weeks the subjects in the TLSO group will decrease and stop the use of the orthesis. Depending on their pain complaints patients will be admitted to the hospital and will get adequate pain management following local protocol Intervention: After fitting the patient starts mobilising, under supervision of a physiotherapist, until pain is under control with oral analgesia. Sports and heavy lifting are prohibited for 3 months. No physiotherapy treatment is needed. During two year follow up patients will be seen at the outpatient clinic during standard care follow up moments. At or just before each scheduled appointment they will fill in questionnaires. These questionnaires will take 15-45 minutes.
  Interventions: Device: Orthesis
- No Orthesis (Active Comparator): Subjects will wear a TLSO for 6 weeks 24 hours a day or they will not. After 6 weeks the subjects in the TLSO group will decrease and stop the use of the orthesis. Depending on their pain complaints patients will be admitted to the hospital and will get adequate pain management following local protocol.
  Control: The patient starts mobilising, under supervision of a physiotherapist, until pain is under control with oral analgesia. Sports and heavy lifting are prohibited for 3 months. No physiotherapy treatment is needed. During two year follow up patients will be seen at the outpatient clinic during standard care follow up moments. At or just before each scheduled appointment they will fill in questionnaires. These questionnaires will take 15-45 minutes.
  Interventions: Behavioral: No orthesis

INTERVENTIONS:
Device: Orthesis
  Other Names: Thoraco-Lumbar-Sacral Orthesis; Hyperextension brace
  Arms: Orthesis
Behavioral: No orthesis
  Other Names: Functional
  Arms: No Orthesis

SUMMARY:
Rationale: Thoracolumbar burst fractures are frequently seen in the trauma population, they have a large impact on patient's wellbeing and are a large economic burden to society. Thoracolumbar burst fractures might not need the standard care of brace immobilization for adequate treatment and a functional treatment might lead to same or better functional outcomes. Besides that, with functional outcome length of hospital stay might decrease and it might also be cost effective compared to bracing.

Objective: The investigators aim to study the use of braces for thoracolumbar burstfractures, not only by measuring the functional scores and the effect of the bracing or functional treatment on the increase in kyphosis angle, but also on (health related) quality of life and health economics. The investigators hypothesize that no treatment is superior over one other.

Study design: This project is a randomised controlled trial comparing brace and no brace treatment on function, kyphosis angle, pain, quality of life, and costs.

Study population: Patients between 18 and 65, with a single level thoracolumbar burst fracture will be included. The fracture has to have a kyphosis angle of less than 35 degrees and patient has to be neurologically intact. Patients are excluded when they are overweight (BMI> 35), need multidisciplinary treatment due to multitrauma, or have inadequate knowledge of the Dutch language. Patients included in the brace group will automatically take part in a brace compliance study.

Intervention: One group receives a Thoracolumbar Sacral Orthesis (TLSO) for 6 weeks, the other group receives no TLSO Main study parameters/endpoints: The primary outcome of this study is the functional score at six months after trauma. Secondary outcomes are pain, kyphosis angle, health related quality of life, healthcare costs and brace compliance.

Literature shows no difference in pain, functional outcome or kyphosis angle, therefore no potential risks are known comparing a brace and a functional treatment. Investigators aim that not using the TLSO results in similar functional outcome, pain and kyphosis angle, and less costs. Patients will be seen at first presentation and during two year follow up at the outpatient clinic at six standard care follow up moments. At these follow up moments a X-ray as part of standard care is made. At or just before each scheduled appointment they will fill in questionnaires taking from 15-45 minutes.

DETAILED DESCRIPTION:
No extra information

ELIGIBILITY:
Inclusion Criteria:

* Th10-L4
* AO foundation type A3 or A4 type fractures
* Single level
* Kyphosis < 35 ° at first analysis
* Neurologically intact
* Adequate trauma

Exclusion Criteria:

* Inadequate knowledge of the Dutch language
* Multitrauma, which asks for multidisciplinary treatment
* Inability to wear a brace due to overweight (BMI> 35)
* Known osteoporosis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Estimated)
Dates: Start 2016-03; Primary Completion 2018-01 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Functional score | at six months, measured up to two years
  Oswestry Disability Index (ODI) derived from the Oswestry Low Back Pain Questionnaire used to quantify disability for low back pain. The self-completed questionnaire contains ten topics concerning intensity of pain, lifting, ability to care for oneself, ability to walk, ability to sit, sexual function, ability to stand, social life, sleep quality, and ability to travel. Each topic category is followed by 6 statements describing different potential scenarios in the patient's life relating to the topic. The patient then checks the statement which most closely resembles their situation. Each question is scored on a scale of 0-5 with the first statement being zero and indicating the least amount of disability and the last statement is scored 5 indicating most severe disability. The scores for all questions answered are summed, then multiplied by two to obtain the index (range 0 to 100). Zero is equated with no disability and 100 is the maximum disability possible.

SECONDARY OUTCOMES:
Quality of life score | up to two years
  WHOQOL-BREF is the short version of the WHOQOL 100 and is recommended for use when time is restricted or the burden on the respondent needs to be minimized. This survey has been used in large epidemiological studies and clinical trials. A self-report questionnaire that contains 26 items and addresses 4 QOL domains: physical health (7), psychological health (6), social relationships (3) and environment (8). Two other items measure overall QOL and general health. Items are rated on a 5-point Likert scale (low score of 1 to high score of 5) to determine a raw item score. Subsequently, the mean score for each domain is calculated, resulting in a mean score per domain that is between 4 and 20. Finally, this mean domain score is then multiplied by 4 in order to transform the domain score into a scaled score, with a higher score indicating a higher QOL. When transformed by multiplying x4, each domain score is then comparable with the scores used in the original WHOQOL-100.
Patient reported health status | up to two years
  The Short Form (SF 36) Health Survey is a 36-item, patient-reported survey of patient health. The SF-36 is a measure of health status and an abbreviated variant of it, the SF-6D, is commonly used in health economics as a variable in the quality-adjusted life year calculation to determine the cost-effectiveness of a health treatment. The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
Quality of life score | up to two years
  The EuroQol-5D is a simple questionnaire with five domains (14). In the EQ-5D, health is defined along five dimensions; mobility, self-care, usual activities, pain or discomfort, and anxiety or depression. Each dimension has three levels; no problem, moderate problem, or severe problem. In addition, a scoring algorithm is available by which each health status description can be expressed into a summary score. This summary score ranges from 1 for full health to 0 for death, and can be interpreted as a judgment on the relative desirability of a health status compared with perfect health.
Pain | up to two years
  Visual Analogue Scale-pain (VAS) is a psychometric response scale which can be used in questionnaires. It is a measurement instrument for subjective characteristics or attitudes that cannot be directly measured. When responding to a VAS item, respondents specify their level of agreement to a statement, in this study pain, by indicating a position along a continuous line between two end-points.
Medical Consumption | up to two years
  The Institute for Medical Technology (iMTA) Medical Consumption Questionnaire (iMCQ), is a generic non disease specific instrument for measuring (direct) medical costs. The instrument is a standardized self-reported questionnaire. The iMCQ includes questions related to frequently occurring contacts with health care providers and can be complemented with extra questions that are relevant for specific study populations. A manual is available for a structured use of the questionnaire. Cost-prices be applied to the obtained healthcare utilization by the iMCQ by using the Dutch manual for cost-analyses that is written by iMTA on behalf of the Dutch Healthcare Institute.
Productivity costs | up to two years
  The Productivity Cost Questionnaire (iPCQ) is a generic non-disease specific questionnaire and is applicable to national and international studies. Currently a Dutch version and an English version of the iPCQ are available. Both indirect cost due to absenteeism as the productivity losses due to presenteeism (i.e. sick, but working) are taken into account. Different methods exist to value productivity. The human-capital method takes the patient's perspective and counts any hour not worked as an hour lost. By contrast, the friction-cost method takes the employer's perspective, and only counts as lost those hours not worked until another employee takes over the patient's work. By applying wage costs the results of the iPCQ can be monetized and as such used in health economic evaluations.
Work Ability | up to two years
  To gain more insight in the effects of a post-trauma status on patients work ability the Work Ability Questionnaire can be used. Originally, the work ability questionnaire consists of 7 dimensions . Recently, it was shown that a very strong association exists between the total Work ability Index (WAI)-score and score on a single-item question (i.e. Current work ability compared with the lifetime best) among all participants. Both the WAI and the single-item question showed similar patterns of associations with sick leave, health, and symptoms. The predictive value for the degree of sick leave and health-related quality of life (HRQoL) was strong for both the WAI and the single-item question. So, it suggests that the single-item question on work ability could be used as a simple indicator for assessing the status and progress of work ability in a working population. Considering the extensive questionnaire being used in the proposed study the single-item questions seems more favourable.

OTHER OUTCOMES:
Length of hospital stay | From first admission until discharge from the hospital up to 10 weeks
  The amount of days spent in the hospital

CONTACTS AND LOCATIONS:
Overall Officials: Taco Gosens, dr., Principal Investigator — Elisabeth Twee Steden ziekenhuis
Locations (1):
- Elisabeth Twee Steden ziekenhuis, Tilburg, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
In this research project the investigators aim for multiple publications in scientific journals and a promotion of a PhD student.
  The investigators want to develop a treating protocol with better functional outcome and less costs.